CLINICAL TRIAL: NCT04218448
Title: Evaluation of the Interest of Hypno-relaxation During Somatosensory Evoked Potentials
Acronym: HYPOT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI's decision
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HYPOT
Record Dates: First submitted 2019-12-30; First posted 2020-01-06 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Neuropathy;Peripheral
MeSH Terms: conditions — Neuritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Somatosensory evoked potentials without hypnorelaxation (No Intervention): As part of this research, the patient must complete a pain scale and a Spielberger Stay-A anxiety self-assessment questionnaire before the PES examination.
  Somatosensory evoked potentials are carried out according to the usual management.
- Somatosensory evoked potentials with hypnorelaxation (Experimental): As part of this research, the patient must complete a pain scale and a Spielberger Stay-A anxiety self-assessment questionnaire before the PES examination. Hypno-relaxation is induced by following VAKOG: external sensory identification, fixation of attention, bodily sensation, breathing, sensory perceptions, closing of the eyes. The work phase follows induction and allows deepening of the hypnotic trance. It corresponds to a metaphorical narrative associated with post-hypnotic suggestions and is fueled by the construction of suggestions and metaphors. The protocol is adapted to each patient. The investigator who remains present throughout the duration of the examination, maintains a hypnotic, empathetic, attentive attitude, and makes it possible to recover this material. The investigator, thanks to hypnosis, allows the development of a creative imagination which allows a modification of the relation to space and time.
  Interventions: Other: Hypnorelaxation

INTERVENTIONS:
Other: Hypnorelaxation — Hypno-relaxation is induced by following VAKOG: external sensory identification, fixation of attention, bodily sensation, breathing, sensory perceptions, closing of the eyes.
  The work phase follows induction and allows deepening of the hypnotic trance. It corresponds to a metaphorical narrative associated with post-hypnotic suggestions and is fueled by the construction of adapted suggestions and metaphors, adapted to each patient. The investigator who remains present throughout the duration of the examination, maintains a hypnotic, empathetic, attentive attitude, and makes it possible to recover this material. Using the elements previously supplied by the patient, the investigator tells a story which allows the patient to focus his attention on something other than the performance of the somatosensory evoked potentials examination. The investigator, thanks to hypnosis, allows the development
  Arms: Somatosensory evoked potentials with hypnorelaxation

SUMMARY:
Somatosensory evoked potentials corresponds to a neurophysiological exam that studies the functioning of the sensitivity pathways. It is often complementary to the imaging examination (MRI or scanner) and the electroneuromyogram which studies only the peripheral part of the sensory and motor pathways while the somatosensory evoked potentials are interested in their central and peripheral component.

The studied information are the potentials generated in the nervous system by the presentation of sensory stimulation. The examination makes it possible to study conduction times which will be defined as normal or pathological according to standards established on control subjects. Their indication is multiple: study of the repercussions of cervical osteoarthritis, specify the diagnosis of certain neuropathies, study of the conduction pathways at the medullary level in the event of trauma or inflammatory or other lesion.

In our study, the investigators will only be interested in the somatosensory evoked Potentials.

A study has shown that hypnotic suggestions to reduce the unpleasantness of pain triggered by thermal stimulation lead to a selective reduction of activity in the anterior cingulate cortex without modifying the activation of the somesthetic cortex.

Pain is, like all sensory stimulation, subject to the influences of attention, anticipation, mental imagery, previous conditioning. The fronto-cingular areas, activated by analgesics such as morphine, or by cortical stimulation are the same as those used by non-drug techniques such as hypnosis.

Therapeutic hypnosis is "a relational experience bringing into play physiological and psychological mechanisms allowing the individual to live better, reduce or eliminate an acute or chronic painful pathology" (Definition of Doctor Jean Marc Benhaiem).

The study of somatosensory evoked Potentials is a long examination (90 to 120 minutes), which can be uncomfortable for the patient (patient lying down, immobile and relaxed), not having to contract his muscles, especially if he is already painful due to his pathology or if it is difficult for him to remain motionless in the supine position. It is indeed necessary to average around 600 to 1000 responses (number of averages) to a small electrical simulation on each member studied.

The muscular contractions of an anxious and/or painful patient prolong the duration of the examination or even disturb the results, to the point of making it impossible to interpret the examination.

To our knowledge, hypnosis has already been used to improve muscle relaxation and reduce anxiety and pain during electromyograms, but hypnosis has never been used to improve the outcome of somatosensory evoked Potentials. Furthermore, if hypnosis modifies certain late cortical waves, it does not cause modification of the early waves and therefore does not disturb the results expected in our clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* Patient who was prescribed PES
* French speaking patient
* Patient affiliated to a social security scheme
* Patient having given oral, free, informed and express consent

Exclusion Criteria:

* Patient with severe pathologies of the peripheral nerve
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Pregnant woman
* Patient denies
* Psychotic patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
duration of the somatosensory evoked potentials | one day
  This correspond to the duration of the somatosensory evoked potentials exam in minuts, between the 2 groups.

SECONDARY OUTCOMES:
Quality of the somatosensory evoked potentials | one day
  This outcome corresponds to the number of averages used to realize the somatosensory evoked potentials exam.

CONTACTS AND LOCATIONS:
Overall Officials: Veronique MARCAUD, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Del Percio C, Triggiani AI, Marzano N, De Rosas M, Valenzano A, Petito A, Bellomo A, Soricelli A, Cibelli G, Babiloni C. Subjects' hypnotizability level affects somatosensory evoked potentials to non-painful and painful stimuli. Clin Neurophysiol. 2013 Jul;124(7):1448-55. doi: 10.1016/j.clinph.2013.02.008. Epub 2013 Apr 25. PMID 23623560
- [Result] Fiorio M, Recchia S, Corra F, Tinazzi M. Behavioral and neurophysiological investigation of the influence of verbal suggestion on tactile perception. Neuroscience. 2014 Jan 31;258:332-9. doi: 10.1016/j.neuroscience.2013.11.033. Epub 2013 Nov 27. PMID 24291728
- [Result] Rainville P, Duncan GH, Price DD, Carrier B, Bushnell MC. Pain affect encoded in human anterior cingulate but not somatosensory cortex. Science. 1997 Aug 15;277(5328):968-71. doi: 10.1126/science.277.5328.968. PMID 9252330
- [Result] Faymonville ME, Laureys S, Degueldre C, DelFiore G, Luxen A, Franck G, Lamy M, Maquet P. Neural mechanisms of antinociceptive effects of hypnosis. Anesthesiology. 2000 May;92(5):1257-67. doi: 10.1097/00000542-200005000-00013. PMID 10781270
- [Result] Lang EV, Benotsch EG, Fick LJ, Lutgendorf S, Berbaum ML, Berbaum KS, Logan H, Spiegel D. Adjunctive non-pharmacological analgesia for invasive medical procedures: a randomised trial. Lancet. 2000 Apr 29;355(9214):1486-90. doi: 10.1016/S0140-6736(00)02162-0. PMID 10801169
- [Result] Stoelb BL, Molton IR, Jensen MP, Patterson DR. THE EFFICACY OF HYPNOTIC ANALGESIA IN ADULTS: A REVIEW OF THE LITERATURE. Contemp Hypn. 2009 Mar 1;26(1):24-39. doi: 10.1002/ch.370. PMID 20161034
- [Result] Vanhaudenhuyse A, Boveroux P, Boly M, Schnakers C, Bruno MA, Kirsch M, Demertzi A, Lamy M, Maquet P, Laureys S, Faymonville ME. [Hypnosis and pain perception]. Rev Med Liege. 2008 May-Jun;63(5-6):424-8. French. PMID 18669215
- [Result] Slack D, Nelson L, Patterson D, Burns S, Hakimi K, Robinson L. The feasibility of hypnotic analgesia in ameliorating pain and anxiety among adults undergoing needle electromyography. Am J Phys Med Rehabil. 2009 Jan;88(1):21-9. doi: 10.1097/PHM.0b013e31818e00bd. PMID 18971768
- [Result] De Pascalis V, Magurano MR, Bellusci A. Pain perception, somatosensory event-related potentials and skin conductance responses to painful stimuli in high, mid, and low hypnotizable subjects: effects of differential pain reduction strategies. Pain. 1999 Dec;83(3):499-508. doi: 10.1016/S0304-3959(99)00157-8. PMID 10568858